CLINICAL TRIAL: NCT05973136
Title: A Pilot Study to Evaluate the Implantation and the Impact of a Hybrid Telerehabilitation Program Based on Cardiopulmonary Rehabilitation Principles for People With Post-COVID Affection
Brief Title: Telerehabilitation for Post COVID-19 Condition
Acronym: Telecovie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Hotel Dieu Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4665
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Long COVID; Chronic Fatigue Syndrome
Keywords: cardiorespiratory; exercise; virtual rehabilitation; post COVID-19 syndrome; fatigue; physiotherapy; post-COVID affection; post-COVID condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic; Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: The study design is a pre-post without a control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Group of participant receiving the hybrid telerehabilitation intervention
  Interventions: Other: Telerehabilitation program based on cardiorespiratory principles

INTERVENTIONS:
Other: Telerehabilitation program based on cardiorespiratory principles — The intervention consists of a hybrid program. The participant will receive rehabilitation sessions in presence (aerobic component of the intervention based on maximal oxygen uptake measured before intervention by means on a ergospirometric test) and at home via a telerehabilitation platform. The length of the intervention is 12 weeks. For the in-presence sessions, they are going to be 75 minutes, 2x/week. For the at-distance sessions, they are going to be 45 minutes, 1x/week in groups of 3 to 4 participants. The intervention will consist of a warm-up, endurance, postural, and strengthening exercises, cool down and respiratory exercises. An exercise book with final recommendations is provided to the participants at the end of the intervention.

SUMMARY:
Telerehabilitation is a great alternative to offering care during a global pandemic. 85% of patients with COVID-19 report persistent symptoms up to 8 months after the infection. There are no clear recommendations for post-covid rehabilitation. The aims of the study are (1) to test the logistic aspect of implanting a hybrid rehabilitation program and (2) to evaluate the acceptability and the potential impact of the program on treating patients with functional limitations and persistent fatigue symptoms. It's a pre and post-study without a control group.

DETAILED DESCRIPTION:
Telerehabilitation is a great alternative to offering care during a global pandemic. 85% of patients with COVID-19 report persistent symptoms up to 8 months after the infection. There are no clear recommendations for post-covid rehabilitation. The aims of the study are (1) to test the logistic aspect of implanting a hybrid rehabilitation program and (2) to evaluate the acceptability and the potential impact of the program on treating patients with functional limitations and persistent fatigue symptoms. It's a pre and post-study without a control group. The intervention will be based on cardiopulmonary rehabilitation principles and will be administered for 12 weeks. Fatigue, post-exertional malaise, and functional/exercise capacities will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Living in the community
* Living near Sherbrooke (<50km)
* Having a diagnostic of COVID-19 confirmed (PCR) and post-COVID syndrome (according to the World Health Organization criteria)
* Being aged between 25 and 65 years old
* Having access to internet at home
* Living with a family member/caregiver or having a telephone or a medical alert system (in case of emergency)
* Reporting persistent fatigue symptoms according to the Fatigue Severity Scale (FSS) (score≥4/7)
* Reporting functional limitations according to the Post-COVID-19 Functional Status scale (PCFS (score ≥2/4);
* Being able to give free and informed consent (adequate understanding of the study protocol);
* Agreeing to perform a pulmonary function test, an exercise stress test, and an ergospirometric exercise test (adequate understanding of steps and procedures);
* Having a low exercise capacity and moderate-to-severe cardiovascular risk <7 metabolic equivalent of a task (MET) or ≤9 if significant reduction of self-reported exercise tolerance according to the stress test performed on a treadmill - Cornell protocol);
* Having no other potential explanatory causes for fatigue or reduced exercise capacity according to medical evaluation

Exclusion Criteria:

* Cognitive impairment: Mini-Mental State Examination (MMSE) ≤24/30
* Inability to perform or understand study procedures
* Medical contraindication

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
The feasibility of the program | 12 weeks
  This will be evaluated by % of participants that accept to participate in the study (recruitment rate), % who completed the intervention (retention rate) and % completed session/anticipated session (adherence).
  The security of the program will be evaluated by the number of falls or near fall.
  Technical difficulty
Acceptability | 12 weeks
  The satisfaction of the participants will be evaluated with a questionnaire (14 questions). The questionnaire will assess patients' satisfaction with the professional, the services and the organization - Telemedicine Satisfaction. Qualitative open-ended questions will be used to determine appreciation and challenges encountered.
Fatigue and post-exercise malaise | 12 weeks
  This will be evaluated with the Fatigue severity scare and De Paul Symptom Questionnaire.

SECONDARY OUTCOMES:
Heart rate variability (resting) | 12 weeks
  Measured with the POLAR H10
Functional capacity | 12 weeks
  Strength, assistance with walking, rising from a chair, climbing stairs, and falls questionnaire (SARC-F)
Exercise capacity | 12 weeks
  6-minute walk test
Lower-limb endurance (estimated) | 12 weeks
  1-minute sit-to-stand test

CONTACTS AND LOCATIONS:
Overall Officials: Livia Pinheiro Carvalho, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada